CLINICAL TRIAL: NCT05956860
Title: Evaluating the Safety and Efficacy of Radial Access for Abdominopelvic Vascular Intervention: a Prospective, Multicenter Study
Brief Title: Radial Access for Abdominopelvic Vascular Intervention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Collaborators: Terumo Medical Corporation (Industry)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: RAVI-202301
Record Dates: First submitted 2023-07-11; First posted 2023-07-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Vascular Access Device Complications
Keywords: Radial access, abdominopelvic vascular intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- radial access for abdominopelvic vascular intervention: abdominopelvic vascular intervention through the radial artery access
  Interventions: Procedure: abdominopelvic vascular intervention through the radial artery access

INTERVENTIONS:
Procedure: abdominopelvic vascular intervention through the radial artery access — According to the pathological changes and needs of the subjects (any abdominal and pelvic arterial intervention that can be performed through the radial artery access, including but not limited to:
  1. hepatic intervention, such as transarterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC), etc.;
  2. Other visceral intervention, such as spleen, kidney, mesentery, etc.;
  3. Pelvic intervention, such as uterine artery embolism, prostatic artery embolism, etc.;
  4. Others, such as preoperative embolization of bone tumors (lumbar, sacral vertebra), etc.

SUMMARY:
To evaluate the safety and efficacy of R.A.V.I.(radial access for abdominopelvic vascular intervention), and evaluate the feasibility and safety of repeated radial artery intervention

DETAILED DESCRIPTION:
This is a prospective, multicenter clinical study with 1143 patients scheduled to enroll based on data from 10 hospitals for any abdominopelvic vascular intervention that can be performed via a radial approach。 The investigators conducted abdominopelvic vascular interventional therapy via radial artery approach according to the lesions and conditions of the subjects.

All subjects underwent Barbeau tests before surgery to examine the flow traffic of the radial and ulnar arteries, and to measure the diameter of the radial artery (inner diameter) by Doppler ultrasound to evaluate its compatibility with the outer diameter of the vascular sheath.

All enrolled subjects were followed up within 24 hours and 1 month after unsheathing to observe the clinical outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. Patients who need abdominopelvic transarterial interventions
3. Preoperative ultrasound assessment of radial artery diameter ≥2mm;
4. Those with good radial pulse and normal Barbeau test (non-D wave);
5. There was no infection, redness swelling or ulceration near the puncture site;
6. Patients and(or) family members agreed to participate in the clinical study and signed informed consent

Exclusion Criteria:

1. Has a history of severe allergy or intolerance to contrast media or chemotherapy drugs;
2. Absence or occlusion of the radial artery pulse;
3. Need large sheath (≥6Fr);
4. Previous history of stroke;
5. Patients with chronic kidney disease who need to establish dialysis access or preserve upper limb blood vessels in the future;
6. Previous history of interventional procedure through radial artery approach (re-intervention of enrolled patients is not included);
7. The investigator believes that the aortic calcification is severe. and the risk of plaque detachment is existed;
8. Patients and(or) family members do not agree to join the clinical trials and sign the informed consent ;
9. According to the investigator's judgment, there are other conditions that are not suitable for participating in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the pathological changes and needs of the subjects (any abdominal and pelvic arterial intervention that can be performed through the radial artery access, including but not limited to:
  1. hepatic intervention, such as transarterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC), etc.;
  2. Other visceral intervention, such as spleen, kidney, mesentery, etc.;
  3. Pelvic intervention, such as uterine artery embolism, prostatic artery embolism, etc.;
  4. Others, such as preoperative embolization of bone tumors (lumbar, sacral vertebra), etc.
Sampling Method: Non-Probability Sample
Enrollment: 1143 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Technical success rate: radial artery puncture success rate and procedure success rate | up to 1 day after surgery
  1)The definition of successful puncture: the radial artery sheath is inserted into the radial artery;
  1. The definition of successful puncture: the radial artery sheath was inserted into the radial artery;
  2. The definition of successful procedure: the catheter was inserted into the target blood vessel via the radial artery, the target procedures was completed, and no crossover to other approach;
Puncture success rate and procedure success rate of repeated radial artery intervention | up to 1 day after surgery
  Repeat radial artery intervention: two or more procedures in the same patient with ipsilateral radial artery intervention.
Complications related to radial approach | up to 1 month after surgery
  a) Minor complications: such as radial artery pulse weakening or disappearance without evidence of distal ischemia, local hematoma* formation or bleeding without blood transfusion or surgical intervention, radial artery spasm*, etc.
  i. Asymptomatic or mild symptoms, no treatment, no sequelae; ii. Minor treatment, including overnight observation only, without sequelae;
  b) Major complication: Such as the need for blood transfusion, limb ischemia, pseudoaneurysm*, any complications requiring surgical intervention, etc.
  i. Short-term hospitalization (<48 hours) ii. Unexpected level of care escalation, prolonged hospital stay(>48 hours) iii. Permanent damage; iv. Die;

SECONDARY OUTCOMES:
Radial artery puncture and sheath insertion time; | up to 1 day after surgery
  The time from the first attempt to puncture with a puncture needle to the successful insertion of the vascular sheath into the radial artery;

OTHER OUTCOMES:
The time of successfully intubation of angiographic catheter; | up to 1 day after surgery
  The time from the angiographic catheter entering the vascular sheath to the first-level branch of the aorta, and the time from the first-level branch of the aorta to the target branch.
Access site crossover rate | up to 1 day after surgery
  The rate of crossing over to the contralateral side through the femoral artery puncture route.
Hemostasis time at the puncture site; | up to 1 day after surgery
  the time from pulling put the sheath to complete hemostasis.
Evaluation of post-procedure comfort | up to 1 month after surgery
  Evaluation of patient comfort using the Post-catheterization Questionaire (1 day after procedure).
Evaluation of post-procedure quality of life | up to 1 month after surgery
  Evaluation of post-procedure quality of life with SF-8 (30 days after procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China